CLINICAL TRIAL: NCT04912739
Title: Targeted Health Dialogues in Primary Care: Lifestyle Screening and Molecular Profiling for a Healthier Life
Brief Title: Targeted Health Dialogues in Primary Care
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02689
Record Dates: First submitted 2021-04-23; First posted 2021-06-03 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Health Behaviors; Risk Factors; Cardiovascular Diseases; Cancer; Serious Diseases
MeSH Terms: conditions — Health Behavior; Cardiovascular Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Targeted health dialogues — Before the targeted health dialogue, the participants fill in a questionnaire about health behaviors, background characteristics and self-rated health. Samples for blood glucose and total cholesterol are taken. BMI, waist-to-hip ratio and blood pressure are measured. The results are summoned in a "health curve", which is discussed with specially trained healthcare personnel in a Targeted heath dialogue. In a sub-group, blood samples are collected for molecular analyses.

SUMMARY:
The County Council of Region Skåne, Sweden, has recently initiated Targeted Health Dialogues in primary care. The prevention program includes health dialogues provided by specially trained personnel, collection of clinical and laboratory data as well as questionnaire data on, e.g., individual health and health behaviors. So far, it enrolls all 40-year old Swedish and foreign-born inhabitants in the county and it will also include all 50- and 60-year old persons within a near future. A research project will be integrated within the program where the collected data will be linked, on the individual level, to national and regional data on hospital admissions, clinical diagnoses from specialist clinics and primary care, causes of death, and prescriptions. The individual linkages will also include population data on sociodemographic characteristics, neighborhood of residence and family relations. Blood samples will be collected for analyses of molecular biomarkers. The research project will examine associations between potential predictors and future risk of cardiovascular diseases and other serious diseases, such as cancer, and also whether the effect of the prevention program is modified by these potential predictors. The effect of the intervention will be examined, and whether the protocol needs to be modified in order to develop more precise and personalized medicine.

DETAILED DESCRIPTION:
The County Council of Region Skåne, the third most populous region in Sweden with 1.4 million inhabitants, has recently initiated Targeted Health Dialogues in primary care with the ultimate goal to improve cardiovascular health in the entire population in Skåne. Targeted health dialogues have previously been proven to improve health behaviors and risk factors and decrease the incidence of cardiovascular disease and mortality. The prevention program includes, in addition to the health dialogues provided by specially trained personnel, collection of clinical and laboratory data (e.g. blood pressure, BMI, waist hip ratio, lipids, fasting blood glucose) as well as detailed questionnaire data on, e.g., individual health and symptoms, family history, diet, physical activity, alcohol and smoking. So far, it enrolls all 40-year old Swedish and foreign-born inhabitants in the county and it will also include all 50- and 60-year old persons within a near future. The County Council and the Ethical Review Board have granted permission to integrate a research project within the program where collected data will be linked, at the individual level, to national and regional data on hospital admissions, clinical diagnoses from specialist clinics and primary care, causes of death, and prescriptions. The individual linkages will also include population data on sociodemographic characteristics, neighborhood of residence and family relations. In addition to the collection and linkages of these data, blood samples will be collected for analyses of molecular biomarkers. The research project will allow for examining associations between a number of potential predictors and future risk of cardiovascular disease and other serious diseases, such as cancer, and also whether the effect of the prevention program is modified by these potential predictors. The effect of the intervention will be examined and whether the protocol needs to be modified in order to develop more precise and personalized medicine.

ELIGIBILITY:
Inclusion Criteria:

* 40-, 50-, 60-, and 70-year old men and women
* Listed at a healthcare center in Skåne county

Exclusion Criteria:

* Inability to understand the written study information and give informed consent

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In Sweden, most people are listed at one healthcare center. The study population consists of all listed 40-, 50-, 60-year, and 70-year-old patients that perform a targeted health dialogue and consent to take part in the research study.
Sampling Method: Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of targeted health dialogues on CVD incidence | 2035
  The short- and long-term effect of targeted health dialogues on incidence of CVD events, its comorbidity and CVD-related deaths in the participants compared to a general population cohort and historical controls.
Effect of targeted health dialogues on incidence of cancer and other serious diseases | 2035
  The short- and long-term effect of targeted health dialogues on incidence of cancer and other serious diseases in the participants compared to a general population cohort and historical controls.

SECONDARY OUTCOMES:
Modification by individual characteristics | 2035
  Modification of possible associations between targeted health dialogues and future CVD, cancer, other serious diseases and preterm death by individual characteristics (e.g., sociodemographic factors)
Association between risk factors and disease incidence | 2035
  Associations between risk factors/combination of risk factors (lifestyle-related, metabolic, psychosocial and familial) at baseline and incidence of CVD, cancer, other serious diseases and preterm death.
Identification of molecular biomarkers | 2035
  The ability of biological aging, epigenetic changes and genetic and metabolomic profiles to predict CVD, cancer, other serious diseases and preterm death as well as the effect of targeted health dialogues.
Public health profile of middle-aged citizens in Sweden's southernmost county | 2035
  Level of physical activity and sedentary behavior, intake of healthy/unhealthy food, alcohol consumption, smoking habits, stress, psychological well-being, blood glucose, cholesterol, BMI, waist-hip ratio. Comparisons between subgroups: age, sex, sociodemography, previous diagnoses.
Associations between dental and general health | 2035
  Associations between dental health at baseline and incidence of CVD, cancer, other serious diseases and preterm death.
Validation of the targeted health dialogue method | 2035
  Validity and reliability of the questionnaire and targeted health dialogue method
Health economy | 2035
  Costs related to the targeted health dialogues versus individual and societal gains.
The effect of targeted health dialogues on health behaviors and self-rated health | 2035
Do targeted health dialogues reach all societal groups? | 2035
Can other lifestyle interventions influence the effect of targeted health dialogues? | 2035
Follow-up of samples taken after the targeted health dialogues. | 2035
  Which samples and tests were taken as a result of the targeted health dialogues?
Do the the targeted health dialogues influence care seeking? | 2035
  Evaluation of new search patterns due to the targeted health dialogues.
Obstacles and motivators for physical activity | 2035
  What obstacles and motivators for physical activity do inactive people experience?
Effect of targeted health dialogues on blood metabolites | 2035
  Do targeted health dialogues affect food-related metabolites in the blood?

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Sundquist, PhD, MD, Principal Investigator — Center for Primary Health Care Research, Department of Clinical Sciences Malmö, Lund University
Locations (1):
- Center for Primary Health Care Research, Lund University and Region Skåne, Malmo, Skåne County, Sweden

REFERENCES:
- [Derived] Nymberg P, Milos-Nymberg V, Grundberg A, Oscarson N, Stenman E, Sundquist K. Exploring the link between self-rated poor oral health and cardiovascular risk: a cross-sectional study using SCORE2. BMC Oral Health. 2025 Feb 24;25(1):298. doi: 10.1186/s12903-025-05671-6. PMID 39994610
- [Derived] Stenman E, Borgstrom Bolmsjo B, Grundberg A, Sundquist K. Health determinants among participants in targeted health dialogues offered to all 40-year-old individuals in a metropolitan region of 1.4 million people. Scand J Prim Health Care. 2025 Mar;43(1):24-35. doi: 10.1080/02813432.2024.2385547. Epub 2024 Aug 1. PMID 39091122